CLINICAL TRIAL: NCT05049785
Title: Nutrition Intervention for Pediatric Patients With Leukemia or Lymphoma Treated With Prednisone and/or Dexamethasone
Brief Title: Nutrition and Physical Activity Intervention in Preventing Excess Weight Gain in Pediatric Patients With Leukemia or Lymphoma Treated With Prednisone and/or Dexamethasone
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2010-0654; NCI-2019-02456 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2010-0654 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-09-09; First posted 2021-09-20 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Leukemia; Lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (counseling) (Active Comparator): Patients attend 13 nutrition counseling sessions over 45 minutes each for 1 year. Patients may receive nutrition handouts.
  Interventions: Other: Counseling; Other: Informational Intervention; Other: Questionnaire Administration
- Arm II (nutrition and PA intervention) (Experimental): Patients attend 2 tasting sessions for low-fat and low-sugar recipes and complete 2 PA sessions over 1 hour for each session.
  Interventions: Behavioral: Exercise Intervention; Dietary Supplement: Nutritional Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Other: Counseling — Attend nutrition counseling sessions
  Other Names: Counseling Intervention
  Arms: Arm I (counseling)
Behavioral: Exercise Intervention — Complete PA sessions
  Arms: Arm II (nutrition and PA intervention)
Other: Informational Intervention — Receive nutrition handouts
  Arms: Arm I (counseling)
Dietary Supplement: Nutritional Intervention — Attend tasting sessions
  Arms: Arm II (nutrition and PA intervention)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies how well a nutrition and physical activity intervention works in preventing excess weight gain in pediatric patients with leukemia or lymphoma treated with Treated with prednisone and/or dexamethasone. A nutrition and physical activity intervention may help develop healthier eating habits and prevent rapid excess weight gain in pediatric patients with leukemia or lymphoma who are receiving prednisone and/or dexamethasone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate if a nutrition counseling intervention will prevent an increase in waist circumference from baseline measurements for children/adolescents diagnosed with leukemia or lymphoma and being treated with prednisone and/or dexamethasone.

SECONDARY OBJECTIVES:

I. To conduct qualitative research on diet habits, likeability of low-fat and-low sucrose foods.

II. To conduct qualitative research on exercise habits and willingness to engage in moderate walking.

III. To assess receptivity to electronic dietary and physical activity (PA) interventions in pediatric cancer patients and survivors (PCPSs) and their parents.

IV. To determine if nutrition interventions will prevent an increase in body mass index (BMI) from baseline measurements for children/adolescents diagnosed with leukemia or lymphoma and being treated with prednisone and/or dexamethasone.

V. To determine if a nutrition counseling intervention will help maintain or decrease triglyceride and cholesterol levels, prevent abnormal values of hemoglobin A1C and improve absolute lymphocyte counts (ALC) from baseline measurements for pediatric leukemia or lymphoma patients, receiving prednisone and/or dexamethasone therapy.

VI. To evaluate caloric intake, nutritional parameters and oxidative stress in pediatric leukemia or lymphoma patients receiving prednisone and/or dexamethasone therapy.

VII. To evaluate responses to various energy balance interventions.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients attend 13 nutrition counseling sessions over 45 minutes each for 1 year. Patients may receive nutrition handouts.

ARM II: Patients attend 2 tasting sessions for low-fat and low-sugar recipes and complete 2 PA sessions over 1 hour for each session.

ELIGIBILITY:
Inclusion Criteria:

* Leukemia or lymphoma patient at MD Anderson Children's Cancer Hospital
* Patients receiving prednisone and/or dexamethasone therapy at MD Anderson Children's Cancer Hospital at time of enrollment
* Karnofsky performance status greater than or equal to 70
* Must be cleared by treating oncologist to participate in study
* Must live close enough to attend measurement sessions at one of the clinical centers

Exclusion Criteria:

* Patients receiving nutrition counseling or weight management counseling elsewhere
* Pediatric patients who are already receiving steroids that are not part of treatment
* History of psychological disorders as indicated in the medical record (eg: eating disorders, depression)

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-05-12 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2025-07-21 (Actual)

PRIMARY OUTCOMES:
Change in waist circumference | through study completion an average of 1 year
  Will assess the difference in waist circumferences between patients in the Arm 1 intervention group compared to patients in the Arm 1 control group. The primary analysis will use the two-sample t-tests, and will be conducted on the intent-to-treat basis. This implies that if patients in the control arm received nutrition counseling, that patient will still be labeled as control.

CONTACTS AND LOCATIONS:
Overall Officials: Joya Chandra, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center website — http://www.mdanderson.org